CLINICAL TRIAL: NCT03455556
Title: Phase I/II Study of the Human Anti-Mesothelin Antibody Drug Conjugate Anetumab Ravtansine (AR), Combined With the PD-L1 Inhibitor Atezolizumab in Non-Small Cell Lung Cancer
Brief Title: Anetumab Ravtansine and Atezolizumab in Treating Participants With Advanced Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1711; NCI-2018-00307 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1711 (Other: Mayo Clinic)
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2020-02

CONDITIONS: Mesothelin Positive; Stage III Non-Small Cell Lung Cancer AJCC v7; Stage IIIA Non-Small Cell Lung Cancer AJCC v7; Stage IIIB Non-Small Cell Lung Cancer AJCC v7; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anetumab ravtansine; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (anetumab ravtansine, atezolizumab) (Experimental): Participants receive anetumab ravtansine IV over 60 minutes and atezolizumab IV over 30-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anetumab Ravtansine; Biological: Atezolizumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Anetumab Ravtansine — Given IV
  Other Names: BAY 94-9343
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the best dose and side effects of anetumab ravtansine when given together with atezolizumab and how well they work in treating participants with non-small cell lung cancer that has spread to other places in the body. Monoclonal antibodies, such as anetumab ravtansine and atezolizumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the recommended phase II dose of anetumab ravtansine combined with atezolizumab in advanced MSLN+ non-small cell lung cancer (NSCLC). (Phase I) II. To determine the confirmed response rate for the combination of anetumab ravtansine and atezolizumab in MSLN+ 2nd line NSCLC. (Phase II)

SECONDARY OBJECTIVES:

I. To describe adverse events and toxicities of the combination treatment of anetumab ravtansine and atezolizumab. (Phase I) II. To identify preliminary evidence of clinical activity (i.e. response, timed endpoints, etc.) (Phase I) III. To determine the progression-free survival (PFS) and the 1-year PFS rate for the combination of anetumab ravtansine and atezolizumab in 2nd-line NSCLC. (Phase II) IV. To determine the overall survival of anetumab ravtansine combined with atezolizumab in second-line therapy of NSCLC. (Phase II) V. Adverse events will also be summarized as well. (Phase II)

CORRELATIVE OBJECTIVES:

I. To determine using flow cytometry the levels of Bcl-2 interacting mediator of cell death (BIM) in circulating CD8+ CD11a+ PD-1+ T-cells, in peripheral blood samples collected from patients prior to initiation of therapy (baseline) and correlating these with confirmed response rate during and following treatment with the combination regimen.

II. To determine tissue MSLN and PD-L1 expression and correlate with response to combination therapy with atezolizumab and anetumab ravtansine.

III. To correlate baseline serum soluble PDL-1 (sPDL-1) with response to therapy.

OUTLINE: This is a phase I, dose-escalation study of anetumab ravtansine followed by a phase II study.

Participants receive anetumab ravtansine intravenously (IV) over 60 minutes and atezolizumab IV over 30-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE REGISTRATION ? INCLUSION CRITERIA: Ability to understand and the willingness to sign a written informed consent document
* PRE REGISTRATION ? INCLUSION CRITERIA: Patient has disease amenable to biopsy if the archival tissue sample is unavailable; note: Archive sample must not be older than 12 months
* REGISTRATION ? INCLUSION CRITERIA
* Phase I only: Diagnosis of advanced/metastatic NSCLC for which no standard treatment option; Phase II only: Advanced NSCLC patients who have received at least 1 platinum-based systemic chemotherapy regimen
* Patients with tumors having actionable genomic alterations should have received prior therapy with Food and Drug Administration (FDA) approved agents targeting these aberrations (ie EGFR, ALK, ROS1, BRAF V600E)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Phase II only: Must have at least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Ability to understand and the willingness to sign a written informed consent document
* Histological or cytologically confirmed NSCLC that shows moderate or stronger mesothelin expression in 30% of tumor cells by a companion assay; MSLN expression score using Ventana immunohistochemistry (IHC) SP74 assay; Phase I only: In addition 5- 30% tumor cells and 1, 2, or 3+ MSLN score; Phase II only: 30% tumor cells and either 2+/3+
* Life expectancy of >= 12 weeks
* Absolute neutrophil count >= 1.5 ? 10^9/L =< 14 days prior to registration
* Platelets >= 100 ? 10^9/L =< 14 days prior to registration
* Hemoglobin >= 9 g/dL =< 14 days prior to registration
* Potassium >= lower limit of normal (LLN) range for the institution =< 14 days prior to registration

  * NOTE: Supplementation may be given before the first dose of study medication
* Calcium >= LLN (corrected for serum albumin, if albumin abnormal) =< 14 days prior to registration

  * NOTE: Supplementation may be given before the first dose of study medication
* Magnesium >= LLN =< 14 days prior to registration

  * NOTE: Supplementation may be given before the first dose of study medication
* Sodium >= LLN =< 14 days prior to registration

  * NOTE: Supplementation may be given before the first dose of study medication
* Phosphorus >= LLN =< 14 days prior to registration

  * NOTE: Supplementation may be given before the first dose of study medication
* International normalized ratio (INR) =< 1.5 =< 14 days prior to registration
* Serum creatinine =< 1.5 mg/dL or creatinine clearance >= 50 mL/min (calculated by Cockcroft Gault equation) =< 14 days prior to registration
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN or =< 5 x upper limits of normal (ULN) if liver metastases are present =< 14 days prior to registration
* Total bilirubin =< 1.5 x ULN =< 14 days prior to registration
* Standard 12-lead electrocardiogram (ECG) with the following parameters at screening (defined as the mean of the triplicate ECGs):

  * QT corrected by Fridericia's formula (QTcF) interval at screening < 450msec (using Fridericia?s correction)
* Negative pregnancy test performed =< 7 days prior to registration (women of childbearing potential only)
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood samples for correlative research purposes

Exclusion Criteria:

* REGISTRATION ? EXCLUSION CRITERIA
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents

  * Note:

    * Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met:

      * Minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose
      * No history of severe immune-related adverse effects from anti-CTLA-4 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] grade 3 and 4)
* More than one prior taxane regimen at any stage of the disease under study (?taxane? refers to paclitaxel, docetaxel, abraxane and cabazitaxel); adjuvant and/or neoadjuvant treatments are considered together as one prior regimen
* Treatment with any other investigational agent or investigational device within 4 weeks prior to registration (or within five half-lives of the investigational product, whichever is longer); patients must be >= 2 weeks since any investigational agent administered as part of a phase 0 study (also referred to as an ?early phase I study? or ?pre phase I study? where a sub- therapeutic dose of drug is administered) at the coordinating center principal investigator (PI)?s discretion, and should have recovered to eligibility levels from any toxicities
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon-alpha or interleukin-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to registration
* Received radiotherapy =< 4 weeks or limited field radiation for palliation =< 2 weeks prior to registration, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom >= 25 percent (%) of the bone marrow was irradiated
* Patients who have a previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study, except

  * Cervical carcinoma in situ, non-melanoma skin cancer, superficial noninvasive bladder tumors, ductal carcinoma in situ (DCIS) or any previous cancer curatively treated >3 years before the start of anetumab ravtansine
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) =< 2 weeks prior to registration

  * Note:

    * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
    * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients with known primary central nervous system (CNS) malignancy or symptomatic CNS metastases are excluded, with the following exceptions

  * Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

    * Evaluable or measurable disease outside the CNS
    * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
    * No history of intracranial hemorrhage or spinal cord hemorrhage
    * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted
    * No neurosurgical resection or brain biopsy =< 28 days prior to registration
  * Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

    * Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
    * No stereotactic radiation or whole-brain radiation =< 28 days prior to registration
    * Screening CNS radiographic study >= 4 weeks from completion of radiotherapy and >= 2 weeks from discontinuation of corticosteroids
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients who have a history or current evidence of bleeding disorder, i.e., any hemorrhage/bleeding event of CTCAE grade >= 2, =< 28 days prior to registration
* History or current evidence of uncontrolled cardiovascular disease including, but not limited to, the following conditions:

  * Congestive heart failure of New York Heart Association (NYHA) class III or IV
  * Unstable angina (symptoms of angina at rest) or new-onset angina =< 6 months before the start of anetumab ravtansine
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with atezolizumab
* Patients on supraphysiologic doses of steroids or use of such =< 6weeks prior to registration
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

  * Note:

    * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener?s granulomatosis, Sjogren?s syndrome, Bell?s palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Note:

    * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible
    * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen are eligible
    * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

      * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
      * Rash must cover less than 10% of body surface area (BSA)
      * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
      * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Severe infections =< 4 weeks prior to registration, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection =< 2 weeks prior to registration
* Major surgical procedure =< 28 days prior to registration or anticipation of need for a major surgical procedure during the course of the study
* Patients with corneal epitheliopathy or any eye disorder that may predispose the patients to this condition as judged by an ophthalmologist

  * Note: Low grades of superficial punctate keratitis, within the range seen in the normal population, should not lead to the exclusion of the patient
* Non-healing serious wound, ulcer, or bone fracture unrelated to the primary tumor
* Previous assignment to treatment during this study; patients permanently withdrawn from study participation will not be allowed to re-enter the study
* Substance abuse, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One (1) patient was recruited from August 2018 to September 2019 at Mayo Clinic. This trial was permanently closed on September 11, 2019. Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Groups:
- Treatment (Anetumab Ravtansine, Atezolizumab): Participants receive 5.5 mg/kg anetumab ravtansine IV over 60 minutes and 1200 mg atezolizumab IV over 30-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Anetumab Ravtansine, Atezolizumab)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Anetumab Ravtansine, Atezolizumab)
Number analyzed (Participants) | 0
Age, Categorical — Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Sex: Female, Male — Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Race (NIH/OMB) — Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Histologic type — Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase I)
Description: Maximum tolerated dose (MTD) of anetumab ravtansine combined with atezolizumab defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients) (Phase I)
Time Frame: Up to 21 days
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Anetumab Ravtansine, Atezolizumab)
Number analyzed (Participants) | 0

2. Primary Outcome: Rate of Confirmed Response (Phase II)
Description: Defined as a patient who has achieved a partial response (PR) or complete response (CR) on two consecutive evaluations at least 4 weeks apart. Will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated.
Time Frame: 6 months
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Anetumab Ravtansine, Atezolizumab)
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinical Activity (Phase I)
Description: Will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population.
Time Frame: Up to 6 months
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Anetumab Ravtansine, Atezolizumab)
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of Adverse Events According to Common Terminology Criteria for Adverse Events Version 4.0 (Phase I)
Description: The number and severity of all adverse events (overall and by dose-level) will be tabulated and summarized in this patient population.
Time Frame: Up to 21 days after last dose
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Anetumab Ravtansine, Atezolizumab)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (Phase II)
Description: Defined as the time from registration to death due to any cause. The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 2 years
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Anetumab Ravtansine, Atezolizumab)
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression-free Survival (Phase II)
Description: Defined as the time from registration to the earliest date of documentation of disease progression or death due to any cause. The distribution of progression-free survival will be estimated using the method of Kaplan Meier. Will also report the 1-year progression free survival (PFS) rate for the combination of anetumab ravtansine and atezolizumab in 2nd-line non-small cell lung cancer (NSCLC).
Time Frame: 1 year and up to 2 years
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Anetumab Ravtansine, Atezolizumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 21 days after last dose
Description: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Anetumab Ravtansine, Atezolizumab)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT03455556/Prot_SAP_000.pdf